CLINICAL TRIAL: NCT06840795
Title: Effect of Vibration Massager Therapy on Non-Specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of Vibration Massager Therapy on Non-Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar20
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): conventional physiotherapy
  Interventions: Other: conventional physiotherapy
- vibration (Experimental): vibration massage therapy in addition to conventional physiotherapy
  Interventions: Other: conventional physiotherapy; Other: Vibration Massage Therapy

INTERVENTIONS:
Other: conventional physiotherapy — Conventional physiotherapy methods will be applied. Pain relief, electrotherapy, hot applications, ultrasound etc.
Other: Vibration Massage Therapy — The device-assisted massage therapy will be applied by the physiotherapist with its gun-shaped form that massages through vibration.
  Arms: vibration

SUMMARY:
The main purpose of this study was to examine the effects of vibratory massage therapy on individuals with non-specific low back pain.

DETAILED DESCRIPTION:
This study will be conducted using a randomized controlled design. Volunteers between the ages of 18-65 with non-specific low back pain will be included in the study. Inclusion criteria are that participants do not have structural pathologies and agree to participate in the study voluntarily. Exclusion criteria include spinal deformities and exercise intolerance. Participants will be randomly divided into two groups. Individuals in the first group will receive vibratory massage therapy, while the second group will be evaluated with standard treatment methods as a control. Both groups will receive treatment 3 times a week for 8 weeks. Participants' quality of life, pain levels, range of motion, and muscle activity will be evaluated before and after treatment. Data will be collected using tools such as SF-36, Oswestry Low Back Pain Index, and VAS (Visual Analog Scale).

ELIGIBILITY:
Inclusion Criteria:

* Having back pain for the last 3 months VAS >4
* Between 18-65 years of age.
* Volunteers for the study.
* Not having undergone surgical intervention in the last 6 months
* Individuals with structural amoli (e.g. spinal deformity).
* Having chronic bone disease

Exclusion Criteria:

* Not being able to cooperate
* Presence of psychological problems
* Use of sleeping pills,
* Presence of neurological and orthopedic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 14 weeks
  The scale is a safe and consistent questionnaire that evaluates the amount of sleep, sleep quality, presence and severity of sleep disorders in individuals in the last month. There are seven components in Pittsburg Sleep Quality Index. These components are subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), sleep medication use (component 6) and daytime dysfunction. (component 7). The evaluation score of each item is between 0-3. The total score obtained varies between 0-21. The higher the score, the worse the sleep quality.
Oswestry Low Back Pain Disability Questionnaire | 14 weeks
  It was developed to measure the functionality of individuals. The scale determines functional disability for activities such as sitting, walking, personal care, lifting, social life, travel, and sleep. There are 10 questions in this scale. Each question has 6 options. Participants are asked to choose the definition that best describes their situation from these options. A score of 0-5 is assigned for each of the sentences, and the highest possible score is 50 points. It is evaluated as mild between 1 and 10 points, moderate between 11 and 30 points, and severe between 31 and 50 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ainaz Vahedi, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lupowitz L. Vibration Therapy - A Clinical Commentary. Int J Sports Phys Ther. 2022 Aug 1;17(6):984-987. doi: 10.26603/001c.36964. eCollection 2022. No abstract available. PMID 36237646
- [Background] Li Q, Liu P, Wang Z, Li X. Vibration therapy to improve pain and function in patients with chronic low back pain: a systematic review and meta-analysis. J Orthop Surg Res. 2023 Sep 26;18(1):727. doi: 10.1186/s13018-023-04217-2. PMID 37752526
- [Background] Leabeater AJ, Clarke AC, James L, Huynh M, Driller M. Under the Gun: Percussive Massage Therapy and Physical and Perceptual Recovery in Active Adults. J Athl Train. 2024 Mar 1;59(3):310-316. doi: 10.4085/1062-6050-0041.23. PMID 37248364
- [Background] Konrad A, Glashuttner C, Reiner MM, Bernsteiner D, Tilp M. The Acute Effects of a Percussive Massage Treatment with a Hypervolt Device on Plantar Flexor Muscles' Range of Motion and Performance. J Sports Sci Med. 2020 Nov 19;19(4):690-694. eCollection 2020 Dec. PMID 33239942